CLINICAL TRIAL: NCT02165566
Title: Humalog or Humulin for Intensive Insulin Therapy in Intensive Care Unit
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Federico Bilotta, Dr, University of Roma La Sapienza
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HlogHlin
Record Dates: First submitted 2014-05-07; First posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Hyperglycemia
Keywords: intensive insulin therapy; critical care patients; blood glucose concentration>180 mg/dl
MeSH Terms: conditions — Hyperglycemia | interventions — Insulin; Insulin, Regular, Human; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regular-insulin, (Experimental): regular-insulin or lispro-insulin at 0.04 units/kg/hour continuous infusion crossover and random assignement
  Interventions: Drug: Regular-insulin
- Lispro insulin (Experimental): patients randomly assigned in a crossover way to one of the 2 treatments
  Interventions: Drug: Lispro-insulin

INTERVENTIONS:
Drug: Regular-insulin — patients are assigned in a random sequence to receive Regular-insulin or lispro-insulin infusion
  Other Names: Humulin
  Arms: Regular-insulin,
Drug: Lispro-insulin — patients are assigned in a random sequence to receive Regular-insulin or lispro-insulin infusion
  Other Names: Humalog
  Arms: Lispro insulin

SUMMARY:
Insulin preparation -random assignment to regular insulin lin or lispro insulin as first treatment- was administered at constant infusion rate (0.04 units/Kg/h) in patients presenting blood glucose concentration ≥180 mg/dl and was discontinued when blood glucose concentration ≤140 mg/dl (therapeutic blood glucose concentration drop). Further reduction in blood glucose concentration after discontinuation of insulin infusion was recorded (post-infusional blood glucose concentration drop). During the study period blood glucose concentration, in whole blood, was measured every 30 minutes. At least 6 hours interval was allowed between the 2 treatments.

DETAILED DESCRIPTION:
Inclusion criteria: Patients older than 18 years of age receiving full nutritional calories supply who presented blood glucose concentration ≥180 mg/dl. Exclusion criteria: moribund patients and patients enrolled on other studies were excluded. Patients with type 1 diabetes, patients with insulin-dependent diabetes are excluded and patients with glycated hemoglobin (glycosilated hemoglobin) >5.6% are also excluded because of the potential of underlying insulin resistance.

A randomized crossover design is used. Patients receiving insulin infusion therapy are prospectively enrolled and randomly assigned to start the treatment either with lispro insulin or regular insulin at a dose of 0.04 units/Kg/h. After full enteral or parenteral nutrition is established, the insulin infusion therapy is started if blood glucose concentration ≥180 mg/dl (upper blood glucose concentration threshold) and is kept constant until blood glucose concentration is ≤140 mg/dl (lower blood glucose concentration threshold). Insulin infusion is discontinued after the blood glucose concentration reached ≤140 mg/dl. Because of the crossover design of the study, the same patient is treated with both lispro insulin or regular insulin infusion allowing an interval of at least 6 hours between the 2 treatments. During the study period -IIT and after insulin infusion is discontinued- the blood glucose concentration is measured every 30 minutes in whole blood (with blood gas analysis) until blood glucose concentration values return within the target threshold (140-180 mg/dl). The primary outcome measure was the extent of "residual effect" after that insulin (Hlog or Hlin) infusion has been discontinued. This variable is expressed as the ratio between blood glucose concentration reduction during insulin infusion (from the beginning of insulin infusion for blood glucose concentration values >180 mg/dl, to the first measurement ≤140 mg/dl) and blood glucose concentration reduction after insulin infusion is discontinued (from the first blood glucose concentration value ≤140 mg/dl to the lowest blood glucose concentration value recorded). Secondary end point measures are: rate of blood glucose concentration reduction during insulin infusion (mg/dl/h-1), duration of the "residual effect" (time elapsed between insulin infusion discontinuation and the lowestblood glucose concentration value), and the rate of blood glucose concentration increase from lowest blood glucose concentration value to the first blood glucose concentration value ≥140 mg/dl.

ELIGIBILITY:
Inclusion Criteria:

* critical care patients with blood glucose concentration >180mg/dl

Exclusion Criteria:

* insulin dependent diabetes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Extent of insulin residual effect in critical care patients | patients will be followed during insulin infusion in a time frame of minutes/hours, with an expected average time of 6-8 hours
  the ratio between the therapeutic effect and the glycemia reduction after insulin is discontinued

CONTACTS AND LOCATIONS:
Overall Officials: Federico Bilotta, MD, PhD, Principal Investigator — Department of Anesthesiology, University of ROme "La Sapienza"
Locations (1):
- University of ROme "La Sapienza" Rome Italy, Rome, Italy

REFERENCES:
- [Derived] Bilotta F, Badenes R, Lolli S, Belda FJ, Einav S, Rosa G. Insulin infusion therapy in critical care patients: regular insulin vs short-acting insulin. A prospective, crossover, randomized, multicenter blind study. J Crit Care. 2015 Apr;30(2):437.e1-6. doi: 10.1016/j.jcrc.2014.10.019. Epub 2014 Oct 30. PMID 25466315